CLINICAL TRIAL: NCT05647122
Title: A Phase I, Multicenter, Open-label, First-in-Human, Dose Escalation and Expansion Study of AZD9592 as Monotherapy and in Combination With Anti-cancer Agents in Patients With Advanced Solid Tumors
Brief Title: First in Human Study of AZD9592 in Solid Tumors
Acronym: EGRET
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D9350C00001; 2022-501570-18-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2022-11-18; First posted 2022-12-12 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumours; Carcinoma Non-small Cell Lung; Head and Neck Neoplasms; Colorectal Neoplasms
Keywords: Cancer; First in Human; Antibody Drug Conjugate; Solid Tumour; Phase I
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Head and Neck Neoplasms; Colorectal Neoplasms; Neoplasms | interventions — osimertinib; Fluorouracil; Leucovorin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Module 1 AZD9592 Monotherapy (Experimental): Module 1 has two parts:
  Part A aims to determine the safety, tolerability, maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D) of AZD9592.
  Part B aims to determine the safety, tolerability and evaluate anti-tumor activity of AZD9592 as monotherapy in select solid tumors
  Interventions: Drug: AZD9592
- Module 2 AZD9592 Combination with Osimertinib (Experimental): Module 2 has two parts:
  Part A aims to determine the safety, tolerability, maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D) of AZD9592 in combination with Osimertinib.
  Part B aims to determine the safety, tolerability and evaluate anti-tumor activity of AZD9592 in combination with Osimertinib in NSCLC EGFRm
  Interventions: Drug: AZD9592; Drug: Osimertinib
- Module 3 AZD9592 Combination 5-FU, Bevacizumab, Leucovorin (Experimental): Module 3 has two parts:
  Part A aims to determine the safety, tolerability and/or recommended phase 2 dose (RP2D) of AZD9592 in combination with 5-FU, Bevacizumab, Leucovorin in Colorectal Cancer (CRC) Part B aims to determine the safety, tolerability and evaluate anti-tumor activity of AZD9592 in combination with 5-FU, Bevacizumab, Leucovorin in Colorectal Cancer (CRC)
  Interventions: Drug: AZD9592; Drug: 5-Fluorouracil (5-FU); Drug: Leucovorin; Drug: Bevacizumab

INTERVENTIONS:
Drug: AZD9592 — Varying doses of AZD9592
Drug: Osimertinib — tablets administered orally
  Arms: Module 2 AZD9592 Combination with Osimertinib
Drug: 5-Fluorouracil (5-FU) — IV infusion
  Arms: Module 3 AZD9592 Combination 5-FU, Bevacizumab, Leucovorin
Drug: Leucovorin — IV infusion
  Arms: Module 3 AZD9592 Combination 5-FU, Bevacizumab, Leucovorin
Drug: Bevacizumab — IV infusion
  Arms: Module 3 AZD9592 Combination 5-FU, Bevacizumab, Leucovorin

SUMMARY:
This is a first-in-human (FIH) Phase I, multi-center, open-label, study of AZD9592, in patients with advanced solid tumors. The study consists of several study modules, each evaluating the safety, tolerability, preliminary efficacy, pharmacokinetics (PK), pharmacodynamics, anti-tumor activity, and immunogenicity of AZD9592, as monotherapy or in combination with anti-cancer agents.

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) Performance Status: 0-1
* Life expectancy ≥ 12 weeks
* Measurable disease per RECIST v1.1
* Adequate organ and marrow function as defined in the protocol

Additional Inclusion Criteria for Module 1:

• Histologically or cytologically confirmed metastatic or locally advanced EGFRmut., NSCLC; metastatic EGFRwt. NSCLC; recurrent or metastatic HNSCC of the oral cavity; metastatic CRC.

Additional Inclusion Criteria for Module 2:

• Histologically or cytologically confirmed metastatic NSCLC EGFRmut.

Additional Inclusion Criteria for Module 3:

• Histologically or cytologically confirmed metastatic CRC.

Key Exclusion Criteria:

* History of (non-infectious) ILD/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
* Spinal cord compression or a history of leptomeningeal carcinomatosis.
* Active infection including tuberculosis and HBV, HCV or HIV
* Brain metastases unless treated (prior treatment required only for Module 1), asymptomatic, stable, and not requiring continuous corticosteroids at a dose of > 10 mg prednisone/day or equivalent for at least 4 weeks prior to start of study treatment.
* Participants with cardiac comorbidities as defined in the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 403 (Estimated)
Dates: Start 2022-12-21 (Actual); Primary Completion 2027-10-06 (Estimated); Study Completion 2027-10-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | From time of Informed Consent to 30 days post last dose of AZD9592
  Number of patients with adverse events by system organ class and preferred term
Incidence of Serious Adverse Events (SAEs) | From time of Informed Consent to 30 days post last dose of AZD9592
  Number of patients with serious adverse events by system organ class and preferred term
Incidence of dose-limiting toxicities (DLT) as defined in the protocol | From time of first dose of AZD9592 to end of DLT period (approximately 21 days)
  Number of patients with at least 1 dose-limiting toxicity (DLT), which is any toxicity defined as a DLT in the Clinical Study Protocol
Incidence of baseline laboratory finding, ECG and vital signs changes | From time of Informed Consent to 30 days post last dose of AZD9592
  measured by laboratory and vital sign variables over time including change from baseline
Proportion of patients with radiological response (ORR) | From date of first dose of AZD9592 up until progression, or the last evaluable assessment in the absence of progression (approximately 2 years)
  Assessed by overall response rate (ORR) defined as the proportion of patients who have a confirmed complete or partial radiological response by the Investigator according to RECIST v1.1 (for patients in the dose expansion cohorts, only)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From date of first dose of AZD9592 up until progression, or the last evaluable assessment in the absence of progression (approximately 2 years)
  The percentage or number of patients with a confirmed investigator assessed complete or partial response according to response criteria in solid tumours (RECIST v1.1)
Duration of Response (DoR) | From date of first dose of AZD9592 up until progression, or the last evaluable assessment in the absence of progression (approximately 2 years)
  The time from date of first response until date of disease progression or last evaluable assessment (RECIST v1.1) in the absence of progression
Disease Control Rate (DCR) at 12 weeks | From date of first dose of AZD9592 up until progression, or the last evaluable assessment in the absence of progression (for each patient this is expected to be measured at 12 weeks)
  The percentage of patients with confirmed CR or PR or having SD maintained (RECIST v1.1) for >=11 weeks from first dose
Progression free Survival (PFS) | From date of first dose of AZD9592 up until date of progression or death due to any cause (approximately 2 years)
  The time from first dose until RECIST 1.1 defined disease progression or death due to any cause
Overall Survival (OS) | From date of first dose of AZD9592 up until the date of death due to any cause (approximately 2 years)
  The time from the date of the first dose of study treatment until death due to any cause.
Pharmacokinetics of AZD9592: Plasma PK concentrations | From date of first dose of AZD9592 up until 30 days post last dose
  Measurement of plasma concentrations of AZD9592, total antibody and total unconjugated warhead
Pharmacokinetics of AZD9592: Area under the concentration time curve (AUC) | From date of first dose of AZD9592 up until 30 days post last dose
  Measurement of PK parameters: Area under the concentration time curve (AUC)
Pharmacokinetics of AZD9592: Maximum plasma concentration of the study drug (C-max) | From date of first dose of AZD9592 up until 30 days post last dose
  Measurement of PK parameters: Maximum observed plasma concentration of the study drug (C-max)
Pharmacokinetics of AZD9592: Time to maximum plasma concentration of the study drug (T-max) | From date of first dose of AZD9592 up until 30 days post last dose
  Measurement of PK parameters: Time to maximum observed plasma concentration of the study drug (T-max)
Pharmacokinetics of AZD9592: Clearance | From date of first dose of AZD9592 up until 30 days post last dose
  Measurement of PK parameters: the volume of plasma from which the study drug is completely removed per unit time (Clearance)
Pharmacokinetics of AZD9592: Half-life | From date of first dose of AZD9592 up until 30 days post last dose
  Measurement of PK parameters: Terminal elimination half-life (t 1/2)
Immunogenicity of AZD9592: Anti-Drug Antibodies (ADA) | From date of first dose of AZD9592 up until 30 days post last dose
  Evaluating the number and percentage of patients who develop Anti-drug antibody (ADA) during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Charu Aggarwal, MD, MPH, Principal Investigator — University of Pennsylvania
Locations (42):
- United States (13):
  - Research Site, Duarte, California
  - Research Site, Irvine, California
  - Research Site, North Haven, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Chicago, Illinois
  - Research Site, Baltimore, Maryland
  - Research Site, Milford, Massachusetts
  - Research Site, Mineola, New York
  - Research Site, New York, New York
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Houston, Texas
  - Research Site, Fairfax, Virginia
- Australia (2):
  - Research Site, Kogarah
  - Research Site, Melbourne
- Canada (2):
  - Research Site, Edmonton, Alberta
  - Research Site, Toronto, Ontario
- China (5):
  - Research Site, Beijing
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Harbin
  - Research Site, Wuhan
- France (3):
  - Research Site, Marseille
  - Research Site, Rennes
  - Research Site, Villejuif
- Italy (4):
  - Research Site, Milan
  - Research Site, Orbassano
  - Research Site, Rozzano
  - Research Site, Verona
- Japan (4):
  - Research Site, Chūōku
  - Research Site, Kashiwa
  - Research Site, Kōtoku
  - Research Site, Osaka
- Malaysia (2):
  - Research Site, Kuala Lumpur
  - Research Site, Kuching
- Research Site, Seoul, South Korea
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Seville
- Taiwan (3):
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home